CLINICAL TRIAL: NCT00956579
Title: MEG/EEG/MRI and Psychophysics Study of Developmental Disorders
Brief Title: Sensory and Connectivity Abnormalities in Autism Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tal Kenet, Associate Professor, Massachusetts General Hospital
Other Study IDs: 2005P001768; 5R01MH117998 (NIH)
Record Dates: First submitted 2007-10-23; First posted 2009-08-11 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; autistic; sensory; MEG; connectivity; brain; MRI; language; developmental; neurodevelopmental; aspergers; asperger's; coherence
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Language

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy individuals: No intervention
  Healthy participants ages 14-32 for a neuroimaging study
- Individuals with Autism Spectrum Disorder: No intervention
  ASD participants ages 14-32 for a neuroimaging study.

SUMMARY:
Study the neural substrates of autism spectrum disorders using neuroimaging methods such as MEG/EEG/MRI.

DETAILED DESCRIPTION:
(NOTE: we are currently recruiting individuals between the ages of 14 and 32, either typically developing or with an autism spectrum disorder.)

To study how sensory information is processed by the brain, we primarily use an instrument called MEG (MagnetoEncephaloGraphy), which measures the magnetic brainwaves emitted by our brains. The device does not have any output (i.e., there is no magnetic field); it only measures the waves produced in the brain.

We measure those waves as the participants in the study listen to, view, or otherwise experience simple, non painful, stimuli. For instance, participants may listen to words while sitting in the MEG room, and watching a movie with the sound turned off.

We then combine this information with pictures of the brain from MRI (Magnetic Resonance Imaging - when available), to get an idea about both the anatomy and the function of the brain, so that we can study how the brains of populations with autism spectrum disorders or language disorders may be different from those of typically developing populations.

ELIGIBILITY:
Inclusion Criteria:

* All of the following criteria must be met by all participants:

  * The participant or the participant's legal guardian is able to understand and is willing to comply with the requirements of the study
  * The participant meets the age requirements (14-32 years old)
  * The participant or legal guardian has signed an Informed Consent Form specific to this study, and is able to understand the consent form.
  * The participant must have English as their first language.
  * The participant must have a non-verbal IQ > 70
* For the ASD/language disorder group only:

  * Autism Spectrum Disorder: Participants must meet criteria for Autism Spectrum Disorder on the ADOS.

Exclusion Criteria:

* The following exclusion criteria apply to both control and autism groups:

  * Any volunteer for whom informed consent cannot be obtained
  * Volunteers with metal braces, extensive dental work involving metals, implanted electromagnetically activated medical equipment (cardiac pacemakers, neurostimulators, functioning infusion pumps), all of which would interfere with the MEG signal, will be excluded from the MEG portion of the study
  * Volunteers with any medically diagnosed sensory loss
  * Volunteers with a known genetic disorder (e.g. Tourette's syndrome, etc), or other medical condition affecting the brain, such as progressive encephalopathy as well as those who are on high doses of multiple anti-seizure medications and have frequent, uncontrolled seizures
  * Asphyxia at birth or any other time, premature birth (Fewer than 34 weeks gestation)
* For the control group only:

  * Volunteers diagnosed with a mental condition such as depression, anxiety, aggression, hyperactivity, attention deficit disorder (with or without hyperactivity).
  * Volunteers who score below the autism spectrum cut-off (in the normal range) on the ADOS and SCQ
  * Volunteers on any sort of neuro-psychopharmacological treatment (including antidepressants, stimulants, antipsychotics, anticonvulsants, benzodiazepines).
* For the autism group only:

  * Children or adults not meeting criteria for autism spectrum disorder
  * Volunteers with co-morbid disorders such as tuberous sclerosis or fragile X.

Ages: 14 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adult/Pediatric
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Saliency of Sensory Stimuli in Developmental Disorders | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tal Kenet, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center or Biomedical Imaging, Charlestown, Massachusetts, United States